CLINICAL TRIAL: NCT00970931
Title: Prevention of Hypertension in Patients With Pre-hypertension: PREVER-prevention Study
Brief Title: Hypertension Prevention in Pre-Hypertensive Individuals
Acronym: PREVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Principal Investigator, Flávio Danni Fuchs, Dr., Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GPPG08621-1
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Pre-hypertension; Hypertension; Cardiovascular Disease
Keywords: hypertension; diuretics
MeSH Terms: conditions — Prehypertension; Hypertension; Cardiovascular Diseases | interventions — Chlorthalidone; Amiloride; Diuretics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- chlortalidone-amiloride (Experimental)
  Interventions: Drug: Chlorthalidone plus amiloride

INTERVENTIONS:
Drug: Chlorthalidone plus amiloride — Oral Chlorthalidone 12.5 mg plus amiloride 2.5 mg, once a day for 18 months
  Other Names: diuretic
  Arms: chlortalidone-amiloride
Drug: placebo — Oral placebo once a day, for 18 months
  Arms: placebo

SUMMARY:
The incidence of hypertension in individuals with pre-hypertension was 80% in ten years in a study conducted in Southern Brazil. The effectiveness of non-drug interventions to prevent hypertension is low in the long term. It may be hypothesized that a population-based drug intervention could reduce relevantly the burden of hypertension and cardiovascular disease.

Diuretics are at least as efficacious as other blood pressure-lowering drugs, are well tolerated, have longer duration of action and the advantage of very low cost to be used in a population intervention. Chlorthalidone is the more efficacious agent. Its main limitation is to induce hypokalemia in a proportion of patients, an adverse effect that can be antagonized by a potassium-sparing diuretic, as amiloride.

A study with this objective is therefore recommendable in Brazil, in order to support a plan of precocious intervention in individuals with pre-hypertension. Such a study was demanded and funded by the Health and Technology Ministries in Brazil.

DETAILED DESCRIPTION:
This is a nation-based trial, with 24 clinical centers distributed in 9 States. A Coordinating Committee is responsible for the elaboration of this proposal and for the main decisions of the trial. The organizational chart of the study will include an executive Committee, a safety committee, outcome committee, lab and EKG centers, and the research units Cardiovascular disease (CVD) is already the leading cause of death in Brazil. High blood pressure is the major risk factor for CVD. The risks start at blood pressure values as lower as 115/75 mmHg but increase exponentially and confer higher absolute risks with blood pressure higher than 140/90 mmHg. The prevalence of hypertension in Brazil was established in population-based studies conducted in different cities and States, varying from 22.3 to 44% of adults The benefit of treatment of individuals with pre-hypertension and cardiovascular disease was demonstrated in several clinical trials. In face of the higher incidence of hypertension in individuals with pre-hypertension, the low effectiveness of non-drug interventions and the risks for cardiovascular events and end-organ damage at lower blood pressure levels, it may be advisable to start blood pressure drugs at low doses at this point of the inexorable elevation of blood pressure with aging.

Research questions

1. Does an association of low doses of chlorthalidone and amiloride reduce the incidence of hypertension in individuals with pre-hypertension?
2. Does an association of low doses of chlorthalidone and amiloride reduce the incidence of cardiovascular events in patients with pre-hypertension?
3. 2. Does an association of low doses of chlorthalidone and amiloride reduce the incidence of target-organ damage in patients with pre-hypertension?

Methods

Design: randomized, double-blind, clinical trial, controlled by placebo.

Eligible participants: individuals with 30 to 70 years of age with pre-hypertension.

Exclusion criteria: low life expectancy, other indications for the use of diuretics, such as cardiovascular disease, intolerance to the study drugs, pregnancy.

Random allocation: by a computer generated list, stratified by center.

Interventions: Chlorthalidone 12.5 mg plus amiloride 2.5 mg or identical placebo.

Primary outcomes:

1. Incidence of hypertension, by blood pressure ≥ 140/90 mmHg in individuals without diabetes or ≥ 135/85 mmHg in participants with diabetes.
2. Adverse events.
3. Development or worsening of microalbuminuria and of left ventricular hypertrophy in the EKG.

ELIGIBILITY:
Inclusion Criteria:

* individuals with 30 to 70 years of age with pre-hypertension

Exclusion Criteria:

* low life expectancy
* other indications for the use of diuretics, such as cardiovascular disease
* intolerance to the study drugs
* pregnancy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2010-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence of hypertension, by blood pressure ≥ 140/90 mmHg in individuals without diabetes or ≥ 135/85 mmHg in participants with diabetes. | 18 months
Adverse events. | 18 months
Development or worsening of microalbuminuria and of left ventricular hypertrophy in the EKG | 18 months

SECONDARY OUTCOMES:
fatal or major cardiovascular events: myocardial infarction, stroke, coronary interventions, heart failure, duplication of creatinine | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Flávio D Fuchs, MD, PhD, Study Chair — Hospital de Clínics de Porto Alegre; Sandra C Fuchs, MD, PhD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Background] Fuchs FD, Fuchs SC, Moreira LB, Gus M, Nobrega AC, Poli-de-Figueiredo CE, Mion D, Bortoloto L, Consolim-Colombo F, Nobre F, Coelho EB, Vilela-Martin JF, Moreno H Jr, Cesarino EJ, Franco R, Brandao AA, de Sousa MR, Ribeiro AL, Jardim PC, Neto AA, Scala LC, Mota M, Chaves H, Alves JG, Filho DC, Pereira e Silva R, Neto JA, Irigoyen MC, Castro I, Steffens AA, Schlatter R, de Mello RB, Mosele F, Ghizzoni F, Berwanger O. Prevention of hypertension in patients with pre-hypertension: protocol for the PREVER-prevention trial. Trials. 2011 Mar 5;12:65. doi: 10.1186/1745-6215-12-65. PMID 21375762
- [Derived] Fuchs FD, Fuchs SC, Poli-de-Figueiredo CE, Figueiredo Neto JA, Scala LCN, Vilela-Martin JF, Moreira LB, Chaves H, Mota Gomes M, de Sousa MR, Silva RPE, Castro I, Cesarino EJ, Sousa ALL, Alves JG, Steffens AA, Brandao AA, Bortolotto LA, Afiune Neto A, Nobrega AC, Franco RS, Sobral Filho DC, Nobre F, Schlatter R, Gus M, De David CN, Rafaelli L, Sesin GP, Berwanger O, Whelton PK. Effectiveness of low-dose diuretics for blood pressure reduction to optimal values in prehypertension: a randomized clinical trial. J Hypertens. 2018 Apr;36(4):933-938. doi: 10.1097/HJH.0000000000001624. PMID 29227377
- [Derived] Fuchs SC, Poli-de-Figueiredo CE, Figueiredo Neto JA, Scala LC, Whelton PK, Mosele F, de Mello RB, Vilela-Martin JF, Moreira LB, Chaves H, Mota Gomes M, de Sousa MR, Silva RP, Castro I, Cesarino EJ, Jardim PC, Alves JG, Steffens AA, Brandao AA, Consolim-Colombo FM, de Alencastro PR, Neto AA, Nobrega AC, Franco RS, Sobral Filho DC, Bordignon A, Nobre F, Schlatter R, Gus M, Fuchs FC, Berwanger O, Fuchs FD. Effectiveness of Chlorthalidone Plus Amiloride for the Prevention of Hypertension: The PREVER-Prevention Randomized Clinical Trial. J Am Heart Assoc. 2016 Dec 13;5(12):e004248. doi: 10.1161/JAHA.116.004248. PMID 27965209